CLINICAL TRIAL: NCT04755881
Title: SHARED (Saguenay Hospitals Anaphylaxis Rule for Early Discharge) - Phase 2 : a Prospective Theoretical Validation
Brief Title: SHARED Study (Saguenay Hospitals Anaphylaxis Rule for Early Discharge)
Acronym: SHARED
Status: Terminated | Type: Observational
Why Stopped: Planned interim data analysis showed underperformance (statistical and clinical) of the three derived clinical decision rules that had been derived and that we were trying to validate.
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Antoine Herman-Lemelin, Principal Investigator, CCFP-ER, MI CPOCUS, Clinical Professor Sherbrooke University, Université de Sherbrooke
Other Study IDs: USherbrooke-SHARED-medfam
Record Dates: First submitted 2021-02-01; First posted 2021-02-16 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Anaphylaxis; Biphasic Anaphylactic Reaction; Rebound Anaphylactic Reaction
Keywords: biphasic anaphylactic reaction; anaphylaxis; allergic reaction; clinical decision rule; anaphylactic reaction; predictors of biphasic anaphylactic reaction; epinephrin; anaphylaxis NIAID/FAAN
MeSH Terms: conditions — Anaphylaxis; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All anaphylaxis reactions seen during the phase 2 period of the SHARED study.: All patients presenting to the 3 sites emergency departments (Chicoutimi, Alma, Jonquière) diagnosed with an anaphylactic reaction or a severe allergic reaction that is rapidly evolving towards anaphylaxis in the opinion of the treating physician.
  Interventions: Other: Occurence of biphasic reaction following anaphylaxis

INTERVENTIONS:
Other: Occurence of biphasic reaction following anaphylaxis — Prospective observation for biphasic reaction following anaphylaxis and subsequent analysis (comparison between usual care and the care that would have been suggested by the three proposed clinical decision rules).

SUMMARY:
Anaphylaxis is a potentially fatal condition with a prevalence between 0.05 and 2% in the general population. This is therefore a frequent reason for emergency visits. Its diagnosis is mainly based on the NIAID / FAAN2 criteria, developed in 2006. The treatment of the condition consists of administration of intramuscular (or intravenous) epinephrine and the hemodynamic support of the patient, if necessary. Various other agents are frequently administered (class I and II antihistamines, corticosteroids) but their role is recognized to be less central than that of epinephrine. The relevance of corticosteroids in reducing the risk of rebound reaction is even questioned.

After anaphylaxis, a serious phenomenon called a "biphasic reaction" can occur. This reaction is the return of symptoms of anaphylaxis resolution of the initial episode. The theoretical risk of a rebound reaction, or biphasic reaction, is conventionally described up to 72 hours after the initial anaphylactic event. Biphasic reaction is defined as a recurrence or occurrence of new signs or symptoms after resolution of the initial reaction, without re-exposure to the allergen. The potential occurrence of a biphasic reaction often warrants observation of patients for several hours in emergency departments following management of the initial anaphylaxis. Although recommendations and guidelines generally suggest observation times of four to six hours, there is no clear consensus or convincing evidence to guide this conduct. It sometimes even is suggested to observe patients for up to 24 hours.

Problem: To date, there are no prognostic factors to identify a patient at greater risk who would benefit from such an observation. As these reactions are a relatively rare phenomenon (i.e. 4 to 5%, but which could go up to 20% according to some sources and the symptoms observed are usually less significant than during the initial presentation, it is therefore possible that a prolonged observation period may not be necessary for some patients who do not have high risk factors for biphasic reaction. In the current context of the growing number of people in emergency rooms and limited ressources, it seems essential to identify low risk patients in order to discharge them quicker and safely by limiting unnecessary observation periods.

Objective: Identify and evaluate in a prospective manner previously derived (literature review and preliminary rules derivation already completed) clinical decision rules that are simple, generalizable and valid which could therefore become an interesting assets for the modern practice of emergency medicine as regards to post anaphylaxis rebound reaction risk stratification. It appears likely that some patients who have suffered an anaphylactic reaction could be safely discharged much earlier than in current practices. The rules would give clear guidelines to clinicians especially those working in lower flow settings, where clinical experience with the disease is less developed. Ultimately, these rules would also be relevant for teaching purposes for the various learners who do internships in emergency rooms.

DETAILED DESCRIPTION:
This study is part of an ongoing projet to create, derive and validate a clinical decision rule with regards to the stratification of the biphasic reaction risk following an anaphylaxis event that has mandated an emergency room visit.

Phase 0: Systematic literature review (completed)

Phase 1: Statistical derivation of two clinical decision rules (retrospective observational study) - (completed)

Phase 2: Validation of clinical decision rules (prospective observational study - theoretical) - (Prematurely terminated)

Objective: The objective of phase 2 was to test the applicability and performance of our clinical decision rules in a prospective observational manner.

UPDATE (March 2023) This unfortunately failed, the rule showed underperformance and clinical utility wasn't attained / maintained in the derivation phase. Furthermore, we tried combining data for the derivation study (phase 1) and the validation study (phase 2) and found that since the phenomenon of biphasic reaction was so heterogeneous, we would need to recruit an unrealistic number of anaphylaxis cases. This endeavor for which we have nor the time, nor the ressources and nor the organizational capabilities would also statistically lead to a clinical decision rule still subject to failure in its further external validations because of the very heterogeneous nature of allergens and the subjects immune reactions to them (projected frailty index).

Methods: Based on the three clinical decision rules (2 derived from phase 1and one based on the literature review), a prospective observational study was carried out in the emergency rooms of Chicoutimi, Jonquière and Alma. Data collection for this theoretical validation phase has been underway since December 2019 and stopped in march 2023, having received the approval of the various local research committees (ethics, science and convenience).

A questionnaire was developed from the three rules derived in the previous phases. All the elements present in these rules have been grouped by categories (history, allergen, symptoms and treatment). In this way, the criteria for each rule were not placed one after the other so that no rule could be recognized or inferred. This questionnaire was presented during department meetings. It is placed on the charts of patients with suspected anaphylaxis at triage and also is available at strategic locations in all three emergency rooms (for example, in the reanimation room).

Doctors were therefore invited to complete the questionnaire anonymously following their initial management of an anaphylactic reaction. Thereafter, they treat the patient as they would have done according to their usual practice. No rules was applied to the patients and the answers provided had no impact on their future care. The questionnaires were then deposited in a secured location determined for this purpose, in each of the emergencies.

The collection of files began in December 2019 and is now terminated. The inclusion and exclusion criteria were the same as in phase 1. However, a patient who did not yet meet the criteria for anaphylaxis, but who, according to the clinician's assessment, would inevitably progress to an anaphylactic reaction could also be included if treated in this way. This was then clearly indicated on the questionnaire.

At the end of the preliminary recruitment period, all completed questionnaire files will be reviewed to determine if a biphasic reaction has occurred. The three clinical decision rules will then be applied to the population to test their performance, validity and safety. The planned interim analysis which led to preliminary termination of the study included 191 cases of anaphylaxis and 11 biphasic reactions (only 6 of which were deemed clinically significant as per protocol criteria).

Some number of anaphylaxis cases were included in the study in between the preliminary analysis (march 2022) and its the results and decision to terminate the study (march 2023). This remaining will of course be analyzed and we propose to publish our data sets in hopes it can be used by other researchers in the field.

Lastly, the investigators were proposing to run a phase 3 trial, if the phase 2 trial had identified valid and clinically usable clinical decision rule(s). That phase 3 trial would have aimed to prospectively validate in real clinical setting and in a different patient population subset the selected rule(s). This phase 3 will unfortunately not be taking place as the trial was prematurely terminated during planned interim analysis in its phase 2 due to clinical uselessness of all 3 rules being tested. Of note, investigators tried to combine data sets from both phases 1 and 2 and still could not derive a rule for which statistical solidity could be expected in the face of such an heterogeneous process as the biphasic allergic reaction is.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages with anaphylaxis (meeting the NIAID/FAAN criteria)
* Patients of all ages considered to be inevitably evolving torwards overt anaphylaxis by the threading physician

Exclusion Criteria:

* Adverse reaction to a medication (eg ACEI)
* Hereditary angioedema
* Known immune mediated Angioedema
* Anaphylactoid reaction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to recruit 533 patients of all ages from three sites of Saguenay-Lac-St-Jean's hospitals' emercgency services (Chicoutimi, Alma and Jonquiere).
  Recruiting started in december 2019 following approval from the ethics comity, sciencitic validity evaluation and institutional convenience.
  Faced with a case of anaphylaxis, the emergency doctor will have to answer a short questionnaire developed with the variables present in each of the three rules.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Rules maintain their sensitivity and negative predictive value with a different sample of patients from the same population pool (prospectively). | December 2019 - 2022
  This phase 2 aims to prospectively verify whether these previously derived or inferred rules maintain their sensitivity and negative predictive value with a different sample of patients from the same population pool. The first rule assesses the probability of clinically significant biphasic reactions (sensitivity of 90% in derivation phase, 7 variables) and the second, all biphasic reactions (sensitivity 100% in derivation phase, 7 variable sensitivity).
  This will allow us to assess the internal validity of the different rules derived from the same three study sites (Chicoutimi, Jonquière, Alma). In addition, the evaluation of the results will help identify the most effective rule.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'urgence CIUSSS du Saguenay - Lac-St-Jean, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Campbell and al., Anaphylaxis: Emergency treatment. UptoDate. 2018
- [Background] Lieberman, P. and al. Biphasic and protracted anaphylaxis. UptoDate. 2018
- [Background] Lieberman P, Nicklas RA, Randolph C, Oppenheimer J, Bernstein D, Bernstein J, Ellis A, Golden DB, Greenberger P, Kemp S, Khan D, Ledford D, Lieberman J, Metcalfe D, Nowak-Wegrzyn A, Sicherer S, Wallace D, Blessing-Moore J, Lang D, Portnoy JM, Schuller D, Spector S, Tilles SA. Anaphylaxis--a practice parameter update 2015. Ann Allergy Asthma Immunol. 2015 Nov;115(5):341-84. doi: 10.1016/j.anai.2015.07.019. No abstract available. PMID 26505932
- [Background] Alqurashi W, Ellis AK. Do Corticosteroids Prevent Biphasic Anaphylaxis? J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1194-1205. doi: 10.1016/j.jaip.2017.05.022. PMID 28888249
- [Background] Simons FE, Ebisawa M, Sanchez-Borges M, Thong BY, Worm M, Tanno LK, Lockey RF, El-Gamal YM, Brown SG, Park HS, Sheikh A. 2015 update of the evidence base: World Allergy Organization anaphylaxis guidelines. World Allergy Organ J. 2015 Oct 28;8(1):32. doi: 10.1186/s40413-015-0080-1. eCollection 2015. PMID 26525001
- [Background] Surveillance report 2016 - Anaphylaxis: assessment and referral after emergency treatment (2011) NICE guideline CG134 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2016 Nov 10. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK551072/ PMID 31855336
- [Background] Brown SG, Stone SF, Fatovich DM, Burrows SA, Holdgate A, Celenza A, Coulson A, Hartnett L, Nagree Y, Cotterell C, Isbister GK. Anaphylaxis: clinical patterns, mediator release, and severity. J Allergy Clin Immunol. 2013 Nov;132(5):1141-1149.e5. doi: 10.1016/j.jaci.2013.06.015. Epub 2013 Aug 1. PMID 23915715
- [Background] Zilberstein J, McCurdy MT, Winters ME. Anaphylaxis. J Emerg Med. 2014 Aug;47(2):182-7. doi: 10.1016/j.jemermed.2014.04.018. Epub 2014 Jun 2. PMID 24881890
- [Background] Campbell RL, Li JT, Nicklas RA, Sadosty AT; Members of the Joint Task Force; Practice Parameter Workgroup. Emergency department diagnosis and treatment of anaphylaxis: a practice parameter. Ann Allergy Asthma Immunol. 2014 Dec;113(6):599-608. doi: 10.1016/j.anai.2014.10.007. No abstract available. PMID 25466802
- [Background] Cheng A. Emergency treatment of anaphylaxis in infants and children. Paediatr Child Health. 2011 Jan;16(1):35-40. PMID 22211074
- [Background] Ring J, Beyer K, Biedermann T, Bircher A, Duda D, Fischer J, Friedrichs F, Fuchs T, Gieler U, Jakob T, Klimek L, Lange L, Merk HF, Niggemann B, Pfaar O, Przybilla B, Ruëff F, Rietschel E, Schnadt S, Seifert R, Sitter H, Varga EM, Worm M, Brockow K. Guideline for acute therapy and management of anaphylaxis: S2 Guideline of the German Society for Allergology and Clinical Immunology (DGAKI), the Association of German Allergologists (AeDA), the Society of Pediatric Allergy and Environmental Medicine (GPA), the German Academy of Allergology and Environmental Medicine (DAAU), the German Professional Association of Pediatricians (BVKJ), the Austrian Society for Allergology and Immunology (ÖGAI), the Swiss Society for Allergy and Immunology (SGAI), the German Society of Anaesthesiology and Intensive Care Medicine (DGAI), the German Society of Pharmacology (DGP), the German Society for Psychosomatic Medicine (DGPM), the German Working Group of Anaphylaxis Training and Education (AGATE) and the patient organization German Allergy and Asthma Association (DAAB). Allergo J Int. 2014;23(3):96-112. doi: 10.1007/s40629-014-0009-1. PMID: 26120521; PMCID: PMC4479483.
- [Background] Simons FE, Ardusso LR, Bilo MB, Cardona V, Ebisawa M, El-Gamal YM, Lieberman P, Lockey RF, Muraro A, Roberts G, Sanchez-Borges M, Sheikh A, Shek LP, Wallace DV, Worm M. International consensus on (ICON) anaphylaxis. World Allergy Organ J. 2014 May 30;7(1):9. doi: 10.1186/1939-4551-7-9. eCollection 2014. PMID 24920969
- [Background] Waserman S, Chad Z, Francoeur MJ, Small P, Stark D, Vander Leek TK, Kaplan A, Kastner M. Management of anaphylaxis in primary care: Canadian expert consensus recommendations. Allergy. 2010 Sep;65(9):1082-92. doi: 10.1111/j.1398-9995.2010.02418.x. Epub 2010 Jun 24. PMID 20584005
- [Background] Muraro A, Roberts G, Simons FE. New visions for anaphylaxis: an iPAC summary and future trends. Pediatr Allergy Immunol. 2008 Aug;19 Suppl 19:40-50. doi: 10.1111/j.1399-3038.2008.00766.x. PMID 18665962
- [Background] Chipps BE. Update in pediatric anaphylaxis: a systematic review. Clin Pediatr (Phila). 2013 May;52(5):451-61. doi: 10.1177/0009922812474683. Epub 2013 Feb 7. PMID 23393309
- [Background] Lee S, Sadosty AT, Campbell RL. Update on biphasic anaphylaxis. Curr Opin Allergy Clin Immunol. 2016 Aug;16(4):346-51. doi: 10.1097/ACI.0000000000000279. PMID 27253484
- [Background] Soar J, Pumphrey R, Cant A, Clarke S, Corbett A, Dawson P, Ewan P, Foex B, Gabbott D, Griffiths M, Hall J, Harper N, Jewkes F, Maconochie I, Mitchell S, Nasser S, Nolan J, Rylance G, Sheikh A, Unsworth DJ, Warrell D; Working Group of the Resuscitation Council (UK). Emergency treatment of anaphylactic reactions--guidelines for healthcare providers. Resuscitation. 2008 May;77(2):157-69. doi: 10.1016/j.resuscitation.2008.02.001. Epub 2008 Mar 20. PMID 18358585
- [Background] Brian H. Rowe; Theodore J. Gaeta. Chapter 14: Anaphylaxis, Allergies, and Angioedema. Tintinalli's Emergency Medicine: A Comprehensive Study Guide, 8e
- [Background] Turner PJ, Jerschow E, Umasunthar T, Lin R, Campbell DE, Boyle RJ. Fatal Anaphylaxis: Mortality Rate and Risk Factors. J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1169-1178. doi: 10.1016/j.jaip.2017.06.031. PMID 28888247
- [Background] Cheng A. Le traitement d'urgence de l'anaphylaxie chez les nourrissons et les enfants. Paediatr Child Health. 2011 Jan;16(1):41-6. No abstract available. French. PMID 22211075
- [Result] Campbell RL, Bashore CJ, Lee S, Bellamkonda VR, Li JT, Hagan JB, Lohse CM, Bellolio MF. Predictors of Repeat Epinephrine Administration for Emergency Department Patients with Anaphylaxis. J Allergy Clin Immunol Pract. 2015 Jul-Aug;3(4):576-84. doi: 10.1016/j.jaip.2015.04.009. Epub 2015 May 29. PMID 26032476
- [Result] Alqurashi W, Stiell I, Chan K, Neto G, Alsadoon A, Wells G. Epidemiology and clinical predictors of biphasic reactions in children with anaphylaxis. Ann Allergy Asthma Immunol. 2015 Sep;115(3):217-223.e2. doi: 10.1016/j.anai.2015.05.013. Epub 2015 Jun 22. PMID 26112147
- [Result] Manivannan V, Hess EP, Bellamkonda VR, Nestler DM, Bellolio MF, Hagan JB, Sunga KL, Decker WW, Li JT, Scanlan-Hanson LN, Vukov SC, Campbell RL. A multifaceted intervention for patients with anaphylaxis increases epinephrine use in adult emergency department. J Allergy Clin Immunol Pract. 2014 May-Jun;2(3):294-9.e1. doi: 10.1016/j.jaip.2013.11.009. Epub 2014 Feb 16. PMID 24811020
- [Result] Confino-Cohen R, Goldberg A. Allergen immunotherapy-induced biphasic systemic reactions: incidence, characteristics, and outcome: a prospective study. Ann Allergy Asthma Immunol. 2010 Jan;104(1):73-8. doi: 10.1016/j.anai.2009.11.001. PMID 20143649
- [Result] Rohacek M, Edenhofer H, Bircher A, Bingisser R. Biphasic anaphylactic reactions: occurrence and mortality. Allergy. 2014 Jun;69(6):791-7. doi: 10.1111/all.12404. Epub 2014 Apr 12. PMID 24725226
- [Result] Pourmand A, Robinson C, Syed W, Mazer-Amirshahi M. Biphasic anaphylaxis: A review of the literature and implications for emergency management. Am J Emerg Med. 2018 Aug;36(8):1480-1485. doi: 10.1016/j.ajem.2018.05.009. Epub 2018 May 9. PMID 29759531
- [Result] Ko BS, Kim WY, Ryoo SM, Ahn S, Sohn CH, Seo DW, Lee YS, Lim KS, Kim TB. Biphasic reactions in patients with anaphylaxis treated with corticosteroids. Ann Allergy Asthma Immunol. 2015 Oct;115(4):312-6. doi: 10.1016/j.anai.2015.07.015. Epub 2015 Aug 12. PMID 26276313
- [Result] Inoue N, Yamamoto A. Clinical evaluation of pediatric anaphylaxis and the necessity for multiple doses of epinephrine. Asia Pac Allergy. 2013 Apr;3(2):106-14. doi: 10.5415/apallergy.2013.3.2.106. Epub 2013 Apr 26. PMID 23667834
- [Result] Mehr S, Liew WK, Tey D, Tang ML. Clinical predictors for biphasic reactions in children presenting with anaphylaxis. Clin Exp Allergy. 2009 Sep;39(9):1390-6. doi: 10.1111/j.1365-2222.2009.03276.x. Epub 2009 May 26. PMID 19486033
- [Result] Grunau BE, Wiens MO, Rowe BH, McKay R, Li J, Yi TW, Stenstrom R, Schellenberg RR, Grafstein E, Scheuermeyer FX. Emergency Department Corticosteroid Use for Allergy or Anaphylaxis Is Not Associated With Decreased Relapses. Ann Emerg Med. 2015 Oct;66(4):381-9. doi: 10.1016/j.annemergmed.2015.03.003. Epub 2015 Mar 25. PMID 25820033
- [Result] Kim TH, Yoon SH, Lee SY, Choi YH, Park CM, Kang HR, Cho SH. Biphasic and protracted anaphylaxis to iodinated contrast media. Eur Radiol. 2018 Mar;28(3):1242-1252. doi: 10.1007/s00330-017-5052-0. Epub 2017 Sep 27. PMID 28956131
- [Result] Jarvinen KM, Amalanayagam S, Shreffler WG, Noone S, Sicherer SH, Sampson HA, Nowak-Wegrzyn A. Epinephrine treatment is infrequent and biphasic reactions are rare in food-induced reactions during oral food challenges in children. J Allergy Clin Immunol. 2009 Dec;124(6):1267-72. doi: 10.1016/j.jaci.2009.10.006. PMID 20004784
- [Result] Kawano T, Scheuermeyer FX, Stenstrom R, Rowe BH, Grafstein E, Grunau B. Epinephrine use in older patients with anaphylaxis: Clinical outcomes and cardiovascular complications. Resuscitation. 2017 Mar;112:53-58. doi: 10.1016/j.resuscitation.2016.12.020. Epub 2017 Jan 6. PMID 28069483
- [Result] Manivannan V, Campbell RL, Bellolio MF, Stead LG, Li JT, Decker WW. Factors associated with repeated use of epinephrine for the treatment of anaphylaxis. Ann Allergy Asthma Immunol. 2009 Nov;103(5):395-400. doi: 10.1016/S1081-1206(10)60358-4. PMID 19927537
- [Result] Reitter M, Petitpain N, Latarche C, Cottin J, Massy N, Demoly P, Gillet P, Mertes PM; French Network of Regional Pharmacovigilance Centres. Fatal anaphylaxis with neuromuscular blocking agents: a risk factor and management analysis. Allergy. 2014 Jul;69(7):954-9. doi: 10.1111/all.12426. Epub 2014 May 10. PMID 24813248
- [Result] Lee S, Peterson A, Lohse CM, Hess EP, Campbell RL. Further Evaluation of Factors That May Predict Biphasic Reactions in Emergency Department Anaphylaxis Patients. J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1295-1301. doi: 10.1016/j.jaip.2017.07.020. PMID 28888253
- [Result] Michelson KA, Monuteaux MC, Neuman MI. Glucocorticoids and Hospital Length of Stay for Children with Anaphylaxis: A Retrospective Study. J Pediatr. 2015 Sep;167(3):719-24.e1-3. doi: 10.1016/j.jpeds.2015.05.033. Epub 2015 Jun 19. PMID 26095285
- [Result] Ellis AK, Day JH. Incidence and characteristics of biphasic anaphylaxis: a prospective evaluation of 103 patients. Ann Allergy Asthma Immunol. 2007 Jan;98(1):64-9. doi: 10.1016/S1081-1206(10)60861-7. PMID 17225722
- [Result] Grunau BE, Li J, Yi TW, Stenstrom R, Grafstein E, Wiens MO, Schellenberg RR, Scheuermeyer FX. Incidence of clinically important biphasic reactions in emergency department patients with allergic reactions or anaphylaxis. Ann Emerg Med. 2014 Jun;63(6):736-44.e2. doi: 10.1016/j.annemergmed.2013.10.017. Epub 2013 Nov 13. PMID 24239340
- [Result] Lee S, Bellolio MF, Hess EP, Campbell RL. Predictors of biphasic reactions in the emergency department for patients with anaphylaxis. J Allergy Clin Immunol Pract. 2014 May-Jun;2(3):281-7. doi: 10.1016/j.jaip.2014.01.012. Epub 2014 Apr 2. PMID 24811018
- [Result] Oya S, Nakamori T, Kinoshita H. Incidence and characteristics of biphasic and protracted anaphylaxis: evaluation of 114 inpatients. Acute Med Surg. 2014 May 19;1(4):228-233. doi: 10.1002/ams2.48. eCollection 2014 Oct. PMID 29930853
- [Result] White JL, Greger KC, Lee S, Kahoud RJ, Li JT, Lohse CM, Campbell RL. Patients Taking beta-Blockers Do Not Require Increased Doses of Epinephrine for Anaphylaxis. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1553-1558.e1. doi: 10.1016/j.jaip.2017.12.020. Epub 2018 Feb 13. PMID 29449164
- [Result] Liyanage CK, Galappatthy P, Seneviratne SL. Corticosteroids in management of anaphylaxis; a systematic review of evidence. Eur Ann Allergy Clin Immunol. 2017 Sep;49(5):196-207. doi: 10.23822/EurAnnACI.1764-1489.15. PMID 28884986
- [Result] Wood JP, Traub SJ, Lipinski C. Safety of epinephrine for anaphylaxis in the emergency setting. World J Emerg Med. 2013;4(4):245-51. doi: 10.5847/wjem.j.issn.1920-8642.2013.04.001. PMID 25215127
- [Result] Dribin TE, Michelson KA, Monuteaux MC, Stack AM, Farbman KS, Schneider LC, Neuman MI. Identification of children with anaphylaxis at low risk of receiving acute inpatient therapies. PLoS One. 2019 Feb 7;14(2):e0211949. doi: 10.1371/journal.pone.0211949. eCollection 2019. PMID 30730977
- [Result] Dribin TE, Michelson KA, Zhang Y, Schnadower D, Neuman MI. Are Children with a History of Asthma More Likely to Have Severe Anaphylactic Reactions? A Retrospective Cohort Study. J Pediatr. 2020 May;220:159-164.e2. doi: 10.1016/j.jpeds.2019.12.019. Epub 2020 Jan 24. PMID 31987654
- [Result] Gabrielli S, Clarke A, Morris J, Eisman H, Gravel J, Enarson P, Chan ES, O'Keefe A, Porter R, Lim R, Yanishevsky Y, Gerdts J, Adatia A, La Vieille S, Zhang X, Ben-Shoshan M. Evaluation of Prehospital Management in a Canadian Emergency Department Anaphylaxis Cohort. J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2232-2238.e3. doi: 10.1016/j.jaip.2019.04.018. Epub 2019 Apr 26. PMID 31035000
- [Result] Kim TH, Yoon SH, Hong H, Kang HR, Cho SH, Lee SY. Duration of Observation for Detecting a Biphasic Reaction in Anaphylaxis: A Meta-Analysis. Int Arch Allergy Immunol. 2019;179(1):31-36. doi: 10.1159/000496092. Epub 2019 Feb 14. PMID 30763927
- [Result] Lee J, Rodio B, Lavelle J, Lewis MO, English R, Hadley S, Molnar J, Jacobstein C, Cianferoni A, Spergel J, Zielinski L, Tsarouhas N, Brown-Whitehorn T. Improving Anaphylaxis Care: The Impact of a Clinical Pathway. Pediatrics. 2018 May;141(5):e20171616. doi: 10.1542/peds.2017-1616. Epub 2018 Apr 3. PMID 29615480
- [Result] Liu X, Lee S, Lohse CM, Hardy CT, Campbell RL. Biphasic Reactions in Emergency Department Anaphylaxis Patients: A Prospective Cohort Study. J Allergy Clin Immunol Pract. 2020 Apr;8(4):1230-1238. doi: 10.1016/j.jaip.2019.10.027. Epub 2019 Nov 6. PMID 31704438
- [Result] Pouessel G, Turner PJ, Worm M, Cardona V, Deschildre A, Beaudouin E, Renaudin JM, Demoly P, Tanno LK. Food-induced fatal anaphylaxis: From epidemiological data to general prevention strategies. Clin Exp Allergy. 2018 Dec;48(12):1584-1593. doi: 10.1111/cea.13287. Epub 2018 Nov 26. PMID 30288817
- [Result] Shaker M, Wallace D, Golden DBK, Oppenheimer J, Greenhawt M. Simulation of Health and Economic Benefits of Extended Observation of Resolved Anaphylaxis. JAMA Netw Open. 2019 Oct 2;2(10):e1913951. doi: 10.1001/jamanetworkopen.2019.13951. PMID 31642933
- [Result] Shaker MS, Wallace DV, Golden DBK, Oppenheimer J, Bernstein JA, Campbell RL, Dinakar C, Ellis A, Greenhawt M, Khan DA, Lang DM, Lang ES, Lieberman JA, Portnoy J, Rank MA, Stukus DR, Wang J; Collaborators, Riblet N, Bobrownicki AMP, Bontrager T, Dusin J, Foley J, Frederick B, Fregene E, Hellerstedt S, Hassan F, Hess K, Horner C, Huntington K, Kasireddy P, Keeler D, Kim B, Lieberman P, Lindhorst E, McEnany F, Milbank J, Murphy H, Pando O, Patel AK, Ratliff N, Rhodes R, Robertson K, Scott H, Snell A, Sullivan R, Trivedi V, Wickham A; Chief Editors, Shaker MS, Wallace DV; Workgroup Contributors, Shaker MS, Wallace DV, Bernstein JA, Campbell RL, Dinakar C, Ellis A, Golden DBK, Greenhawt M, Lieberman JA, Rank MA, Stukus DR, Wang J; Joint Task Force on Practice Parameters Reviewers, Shaker MS, Wallace DV, Golden DBK, Bernstein JA, Dinakar C, Ellis A, Greenhawt M, Horner C, Khan DA, Lieberman JA, Oppenheimer J, Rank MA, Shaker MS, Stukus DR, Wang J. Anaphylaxis-a 2020 practice parameter update, systematic review, and Grading of Recommendations, Assessment, Development and Evaluation (GRADE) analysis. J Allergy Clin Immunol. 2020 Apr;145(4):1082-1123. doi: 10.1016/j.jaci.2020.01.017. Epub 2020 Jan 28. PMID: 32001253.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04755881/Prot_SAP_000.pdf